CLINICAL TRIAL: NCT02542657
Title: Phase I/II Study of Ixazomib in Combination with Pomalidomide, Clarithromycin and Dexamethasone (PiC-D) in Patients with Double Refractory Multiple Myeloma
Brief Title: Ixazomib with Pomalidomide, Clarithromycin and Dexamethasone in Treating Patients with Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Joseph Tuscano (Other)
Collaborators: Takeda (Industry); Celgene (Industry)
Responsible Party: Sponsor-Investigator, Joseph Tuscano, Principal Investigator, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 728937; UCDCC#253 (Other: UC Davis); X16043 (Other Grant/Funding Number: Takeda); UCDCC#253 (Other: University of California Davis Comprehensive Cancer Center); PO-TR-MM-PI-004614 (Other Grant/Funding Number: Celgene)
Record Dates: First submitted 2015-05-08; First posted 2015-09-07 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Myeloma
MeSH Terms: conditions — Neoplasms, Plasma Cell | interventions — Clarithromycin; Dexamethasone; Calcium Dobesilate; ixazomib; pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (PiC-D therapy) (Experimental): Patients receive pomalidomide PO QD on days 1-21; ixazomib citrate PO on days 1, 8, and 15; clarithromycin PO BID on days 15-21 of course 1 and days 1-21 of courses 2-6; and dexamethasone PO on days 1, 8, 15, and 22. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY:
  Patients receive pomalidomide, ixazomib citrate, and dexamethasone as above and receive clarithromycin PO BID or QD. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Clarithromycin; Drug: Dexamethasone; Drug: Ixazomib Citrate; Drug: Pomalidomide

INTERVENTIONS:
Drug: Clarithromycin — Given PO
  Other Names: Biaxin
Drug: Dexamethasone — Given PO
  Other Names: Decadron
Drug: Ixazomib Citrate — Given PO
  Other Names: MLN9708
Drug: Pomalidomide — Given PO
  Other Names: Pomalyst

SUMMARY:
This phase I/II trial studies the side effects and best dose of clarithromycin when given together with ixazomib citrate, pomalidomide, and dexamethasone and to see how well it works in treating patients with multiple myeloma that has not responded to previous treatment. Biological therapies, such as clarithromycin, pomalidomide, and dexamethasone, use substances made from living organisms that may stimulate the immune system in different ways and stop cancer cells from growing. Ixazomib citrate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving clarithromycin with ixazomib citrate, pomalidomide and dexamethasone may be a better treatment for patients with multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the maximum tolerated dose (MTD) and the recommended phase 2 dose (RP2D) for PiC-D therapy (pomalidomide, ixazomib [ixazomib citrate], clarithromycin, and dexamethasone) in patients with multiple myeloma who are bortezomib and lenalidomide refractory. (Phase I) II. To determine the complete response (CR) and stringent CR (sCR) rate for PiC-D therapy in patients with multiple myeloma who are bortezomib and lenalidomide refractory. (Phase II)

SECONDARY OBJECTIVES:

I. To evaluate the safety and tolerability of PiC-D therapy. (Phase I) II. To characterize the pharmacokinetics (PK) in plasma of oral ixazomib in combination with pomalidomide, clarithromycin and dexamethasone. (Phase I) III. To assess preliminary evidence of clinical activity. (Phase I) IV. To assess the effects of PiC-D therapy on quality of life (QOL). (Phase I) V. To assess the effects of PiC-D therapy on immune status (phenotypic analysis and cytokine profiling).

VI. To evaluate the safety of PiC-D therapy. (Phase II) VII. To determine the overall response rate (ORR) (ORR; CR, sCR, partial response, and very good partial response. (Phase II) VIII. To determine the clinical benefit rate (CBR) (CBR; minimal response + ORR). (Phase II) IX. To determine the disease control rate (DCR) (DCR; stable disease + CBR). (Phase II) X. To determine the duration of response (DOR) in patients achieving a partial response or better. (Phase II) XI. To determine the time to next treatment (TNT). (Phase II) XII. To determine progression free survival (PFS) and overall survival (OS). (Phase II) XIII. To assess the effects of PiC-D therapy on quality of life (QOL). (Phase II)

TERTIARY OBJECTIVES:

I. To assess the effects of PiC-D therapy on immune status (phenotypic analysis and cytokine profiling). (Phase II)

OUTLINE: This is a phase I, dose-escalation study of clarithromycin followed by a phase II study.

Patients receive pomalidomide orally (PO) once daily (QD) on days 1-21; ixazomib citrate PO on days 1, 8, and 15; clarithromycin PO twice daily (BID) on days 15-21 of course 1 and days 1-21 and courses 2-6; and dexamethasone PO on days 1, 8, 15, and 22. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY:

Patients receive pomalidomide, ixazomib citrate, and dexamethasone as above and receive clarithromycin PO BID or QD. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 2-3 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written consent
* Patients must have a confirmed biopsy diagnosis of a multiple myeloma
* Submission of original biopsy for review and verification by hematopathologist at local institution
* Patients must have measurable disease according to International Myeloma Working Group (IMWG) criteria; measurable disease includes at least one of the following criteria:

  * Serum M-protein >= 1.0 g/dL, and/or
  * Urine M-protein >= 200 mg/24 hours, and/or
  * Involved serum free light chain >= 10 mg/dL (>= 100 mg/L) AND an abnormal serum free light chain ratio, and/or
  * Baseline marrow burden or myeloma of at least 30%
* Disease that has progressed during or within 6 months of coming off therapy with bortezomib and lenalidomide (either sequentially or concurrent); progressive disease is defined as any of the following:

  * An increase of >= 25% from lowest response value in any of the following:

    * Serum M-protein (absolute increase must be >= 0.5 g/dL) AND/OR
    * Urine M-protein (absolute increase must be >= 200 mg/24 hours) AND/OR
    * For patients without a measurable serum or urine M-protein but measurable disease by serum free light chain testing: Difference between the involved and uninvolved serum free light chain level (absolute increase must be >= 10 mg/dL) AND/OR
    * For patients without a measurable serum or urine M-component or serum free light chain level: % marrow involvement with myeloma (absolute increase must be >= 10%) AND/OR
  * Definite development of new bone lesions or extramedullary plasmacytomas or definite increase in the size of existing bone lesions or extramedullary plasmacytomas AND/OR
  * Hypercalcemia (corrected serum calcium > 11.5 mg/dL) attributable to myeloma (e.g. not due to omitted doses of bisphosphonate)
* Life expectancy of greater than 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status and/or other performance status 0, 1, or 2
* Disease free of prior malignancies for > 5 years with exception of patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection
* Absolute neutrophil count (ANC) >= 1,000/mm^3 and
* Platelet count >= 50,000/mm^3; note: platelet transfusions to help patients meet eligibility criteria are not allowed within 3 days before study enrollment
* Total bilirubin =< 2.0 × the upper limit of the normal range (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 × ULN
* Calculated creatinine clearance >= 30 mL/min
* Female patients who:

  * Are postmenopausal for at least 1 year before the screening visit, OR
  * Are surgically sterile, OR
  * If they are of childbearing potential, agree to practice two effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject (periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception)
* Male patients, even if surgically sterilized (i.e., status post-vasectomy), must agree to one of the following:

  * Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject; (periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception)

Exclusion Criteria:

* Female patients who are lactating or have a positive serum pregnancy test during the screening period
* Treatment with clarithromycin, anti-myeloma therapy including investigational agents or plasmapheresis within 30 days prior to treatment in this study
* Failure to have fully recovered (i.e., =< grade 1 toxicity or to patient's clinical baseline) from the reversible effects of prior chemotherapy
* Major surgery within 14 days before enrollment
* Radiotherapy within 14 days before enrollment
* Central nervous system involvement
* Infection requiring systemic antibiotic therapy or other serious infection within 14 days before study enrollment
* Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months
* Systemic treatment within 14 days before the first dose of study drugs, or concurrent use, with any of the following:

  * Strong inhibitors of cytochrome P450, family 1, subfamily A, polypeptide 2 (CYP1A2)
  * Strong inhibitors of family cytochrome P450 family 3, subfamily A (3A)
  * Strong cytochrome 3A polypeptide 4 inducers
* Known ongoing or active systemic infection, active hepatitis B or C virus infection
* Patients with human immunodeficiency virus (HIV) infection may be eligible provided they meet the following:

  * No history of acquired immunodeficiency syndrome (AIDS)-defining conditions or other HIV related illness
  * Cluster of differentiation (CD)4+ cells nadirs > 350/mm^3
  * Treatment sensitive HIV and, if on anti-HIV therapy, HIV viral load < 50 copies/mm^3; please note: HIV+ patients who enroll on this study may need to modify their anti-retroviral therapy prior to receiving protocol therapy if they are on strong inducers or potent inhibitors of cytochrome P450; adverse events in HIV+ patients will be reported separately
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent
* Previous allergic reaction to an immunomodulatory drug (IMiD)
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of study drugs including difficulty swallowing
* Patient has >= grade 3 peripheral neuropathy, or grade 2 with pain on clinical examination during the screening period
* Previous treatment with ixazomib or pomalidomide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-10; Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
MTD of clarithromycin when given in combination with ixazomib citrate, pomalidomide, and dexamethasone assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 (Phase I) | 28 days
  The MTD is defined as the highest dose tested in which fewer than 33% of patients experience a dose limiting toxicity and at least 6 patients have been treated at that dose. The MTD will be the recommended Phase 2 dose, provided that other safety considerations are acceptable.

SECONDARY OUTCOMES:
Clinical best response | Up to 3 years
  Will be listed for each patient and summarized using standard descriptive methods.

OTHER OUTCOMES:
Change in immune modulation with the addition of clarithromycin (Phase II) | Up to 3 years
  Regression methods (adapted for repeated measures) will be used to describe the changes over time; these regression models will contain contrasts to compare changes from baseline to day 15, and from day 1 of subsequent cycles. P-values calculated based on the regression analyses will be used to calibrate the strength of associations and patterns observed, rather than for drawing definitive conclusions. Additional analysis will be undertaken to explore the relationship between changes (or lack of changes) and response.
Change in immune modulation without the addition of clarithromycin (Phase II) | Baseline to up to 3 years
  Regression methods (adapted for repeated measures) will be used to describe the changes over time; these regression models will contain contrasts to compare changes from baseline to day 15, and from day 1 of subsequent cycles. P-values calculated based on the regression analyses will be used to calibrate the strength of associations and patterns observed, rather than for drawing definitive conclusions. Additional analysis will be undertaken to explore the relationship between changes (or lack of changes) and response.
Pharmacokinetic parameters of ixazomib citrate (Individual and mean plasma ixazomib concentration data) | At 0.5, 1, 1.5, 2, 4, 8, and 24 hours after ixazomib citrate administration on days 1 and 8
  Individual and mean plasma ixazomib concentration data will be plotted over time. A summary table will be presented for the plasma concentration data.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Tuscano, Principal Investigator — University of California, Davis
Locations (3):
- United States (3):
  - University of California San Diego, La Jolla, California
  - University of California Irvine, Orange, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rosenberg AS, Maverakis E, Costello C, Brem EA, Wieduwilt MJ, Luxardi G, Kaesberg P, Abedi K, Herbert S, Tuscano J. Clarithromycin, ixazomib, pomalidomide, dexamethasone for relapsed/refractory myeloma: survival and correlative analysis. Blood Neoplasia. 2025 Jan 16;2(3):100067. doi: 10.1016/j.bneo.2025.100067. eCollection 2025 Aug. PMID 40948663